CLINICAL TRIAL: NCT05760859
Title: Effects of Initial Cues and the Quality of Medical History Taking on Diagnostic Accuracy
Brief Title: Quality of Medical History Taking and Diagnostic Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4031_Sim_MedHistory
Record Dates: First submitted 2023-02-20; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Diagnostic Error
Keywords: medical simulation; diagnostic error; pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Participants were randomized (computer-generated numbers) to six versions of a simulated scenario of pulmonary embolism. The six versions differed only in the initial cues, i.e. in the reply of the patient to the initial question about the reason for his visit.
Who Masked: Participant
Masking Description: Single-blind trial; participants not aware of the goal of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Chest pain (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Chest pain"
  Interventions: Other: Initial cue
- Dyspnoea (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Dyspnoea"
  Interventions: Other: Initial cue
- Chest pain AND Dyspnoea (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Chest pain, and Dyspnoea"
  Interventions: Other: Initial cue
- Chest pain AND dyspnoea, AND leg pain (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Chest pain, and Dyspnoea, and leg pain"
  Interventions: Other: Initial cue
- Chest pain AND dyspnoea, AND immobilization (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Chest pain, and Dyspnoea, and immobilization"
  Interventions: Other: Initial cue
- Chest pain AND dyspnoea, AND leg pain AND immobilization (Experimental): Patient answers the initial question of history taking on why he had come to the hospital with "Chest pain, and Dyspnoea, and leg pain, and immobilization"
  Interventions: Other: Initial cue

INTERVENTIONS:
Other: Initial cue — Symptom volunteered by the "patient"

SUMMARY:
This prospective randomized simulator-based single-blind trial aimed to investigate the effects of initial cues and history taking skills on diagnostic accuracy

DETAILED DESCRIPTION:
Diagnostic errors are a relevant health-care problem. As medical history taking is usually the first step in a patient's assessment its quality is most likely a first and important barrier against diagnostic errors. There are, however, only limited data on the association of the quality of medical history taking and diagnostic accuracy.This prospective randomized simulator-based single-blind trial aimed to investigate the effects of initial cues and history taking skills on diagnostic accuracy. 198 medical students (135 females) were given the task to assess a patient presenting with simulated acute pulmonary embolism. Participants were randomized to six versions of the scenario differing only in the initial cues, i.e. in the reply of the patient to the initial question about the reason for his visit. In three of six versions, initial cues were restricted to thoracic symptoms (chest pain, dyspnoea, or combination of both). In the remaining three versions, initial cues consisted of thoracic and extra-thoracic (leg pain, immobilization) symptoms. The primary outcome was diagnostic accuracy. The mannequin was equipped with a speaker in its head that broadcasts the voice of a remote operator (experienced physician) allowing verbal interaction of the participants with the "patient". The "patient" did not speak unless asked and responded to all participants' questions during history taking according to a pre-defined checklist.

ELIGIBILITY:
Inclusion Criteria:

* 4th year medical students participating in voluntary simulator-based workshops

Exclusion Criteria:

* decline to give written informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Stating the correct diagnosis | 5 minutes
  At the end of the study time (5 minutes), a study physician enters the simulator room and asks the participate on his/her presumptive diagnosis. Simualtions are video-taped and the analysis of the outcome is performed by trained observers by video analysis. "Stating the correct diagnosis" is a binary outcome, rated either as "yes" (correct presumptive diagnosis of pulmonary embolism is stated) or "no" (correct presumptive diagnosis of pulmonary embolism is NOT stated).

SECONDARY OUTCOMES:
Depth of history taking | 5 minutes
  Data analysis is performed using video-recordings recorded during scenarios. Trained observers note kind and timing of all questions. Questions were categorized in six pre-defined categories (chest pain, dyspnoea,associated symptoms, risk factors for pulmonary embolism,cardiovascular risk factors, personal history). Depth of information gathering is assessed for each category separately and is defined as the total number of questions asked in any given category.
Breadth of history taking | 5 minutes
  Data analysis is performed using video-recordings recorded during scenarios. Trained observers note kind and timing of all questions. The three problem areas chest pain, dyspnea, and leg pain or leg swelling were defined à priori as relevant. Breadth of information gathering is defined as number of relevant problem areas identified (possible range from 0 to 3).
Systematics of history taking | 5 minutes
  Data analysis is performed using video-recordings recorded during scenarios. Trained observers note kind and timing of all questions. Questions were categorized in six pre-defined categories (chest pain, dyspnoea,associated symptoms, risk factors for pulmonary embolism,cardiovascular risk factors, personal history). All questions will be rated as either "systematic question" or "non-systematic question". A systematic questions is defined as question, that is either immediately preceded or immediately followed by a question of the same category. "Systematic questions" will be expressed as percentage of all questions asked during history taking (possible range 0% to 100%)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Marsch, MD, Principal Investigator — University Hospital of Basel
Locations (1):
- University Hospital, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
Video recordings are confidential and cannot be shared. Extracted data can be shared upon reasonable request